CLINICAL TRIAL: NCT03490760
Title: Phase II Trial of In Situ Tumor Vaccination Using Durvalumab and "Booster" Radiation Therapy in Patients With Metastatic Adenocarcinoma of the Pancreas Who Have Progressed Through First-line Chemotherapy
Brief Title: Durvalumab and "Booster" Radiation in Metastatic Adenocarcinoma of the Pancreas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow/poor enrollment
Sponsor: Baptist Health South Florida (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR 15 11078
Record Dates: First submitted 2018-03-14; First posted 2018-04-06 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Adenocarcinoma of the Pancreas
Keywords: Metastatic Adenocarcinoma of the Pancreas
MeSH Terms: interventions — durvalumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Single-arm Phase II
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab plus Radiation Therapy (Experimental): Durvalumab 1500 mg (or 20 mg/m2 if <30 kg) IV every 4 weeks plus 24 Gy in 3 daily fractions to one lesion during Week 3 and 24 Gy in 3 daily fractions to the second lesion during Week 5.
  Interventions: Drug: Durvalumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500 mg (or 20 mg/m2 if <30 kg) IV every 4 weeks
Radiation: Radiation Therapy — 24 Gy in 3 daily fractions to one lesion during Week 3 and 24 Gy in 3 daily fractions to the second lesion during Week 5.

SUMMARY:
This is a single-institution, single-arm phase II trial of Durvalumab combined with Radiation Therapy (RT) for metastatic pancreatic cancer patients who have progressed through first-line chemotherapy.

DETAILED DESCRIPTION:
This is a single-institution phase II trial of Durvalumab combined with Radiation Therapy (RT) for metastatic pancreatic cancer patients who have progressed through first-line chemotherapy. Pancreatic cancer patients who have received second-line or greater chemotherapy in the metastatic setting are not eligible. Target accrual is 39 patients. Durvalumab 1500 mg (or 20 mg/m2 if <30 kg) IV every 4 weeks will be started and continued during RT and afterwards until the patient experiences either unacceptable toxicity or disease progression, whichever comes first. Patients must have at least three radiographically measurable pancreatic cancer lesions in different organs that have not previously received RT, two of which will receive RT. Eligible lesions include either the primary pancreatic tumor in unresected patients or distant metastatic lesions. Three fractions of 8 Gy each will be prescribed to one lesion during Week 3. Three fractions of 8 Gy each will be prescribed to the second lesion during Week 5.

This is a single-arm trial with continuous monitoring of acute non-hematologic toxicity with the primary endpoint of progression free survival. Efficacy will be evaluated by time to progression or death, whichever comes first, and compared to historical control of chemotherapy alone as reported in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven metastatic pancreatic adenocarcinoma with progression through standard first-line chemotherapy. Chemotherapy given as part of prior chemoradiation does not count as a line of therapy. Chemotherapy given as part of prior chemoradiation in the setting of non-metastatic pancreatic cancer does not count as a line of therapy.
* At least 3 radiographically distinct pancreatic cancer lesions that are measurable by RECIST 1.1 criteria, including 2 that are eligible for RT.
* Lesions that will receive RT are separated by ≥3 cm and none >7 cm in greatest dimension.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of ≥12 weeks.
* Adequate liver and kidney function.
* Adequate blood cell count.
* Female subjects must either be of non-reproductive potential or must have a negative serum pregnancy test upon study entry.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study
* Previous enrollment in the present study.
* Any previous treatment with a programmed cell death 1 or programmed cell death ligand 1 inhibitor including Durvalumab.
* Prior RT to any lesion that would receive RT on this protocol.
* Prior RT that could lead to an unacceptably high risk of clinically significant normal tissue injury due to high cumulative normal tissue dose as determined by the investigator.
* Subjects who have received more than 1 line of chemotherapy in the metastatic setting.
* History of another primary malignancy except for: 1) malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence; 2) adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; 3) adequately treated carcinoma in situ without evidence of disease (e.g., cervical cancer in situ).
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤14 days prior to the first dose of study drug.
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of Durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Any unresolved toxicity (> grade 2, Common Terminology Criteria for Adverse Events version 4.03) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy).
* Any prior Grade ≥ 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved immune-related adverse event (irAE) >Grade 1.
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Graves' disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency.
* History of allogeneic organ transplant.
* History of liver cirrhosis and Child-Pugh class B or C.
* History of hypersensitivity to Durvalumab or any excipient.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Known history of previous clinical diagnosis of tuberculosis
* History of leptomeningeal carcinomatosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.
* Subjects with uncontrolled seizures.
* Subjects with known radiation hypersensitivity syndromes such as Ataxia-Telangiectasia or Nijmegen Breakage Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Chuong, MD, Principal Investigator — Miami Cancer Institute at Baptist Health, Inc.
Locations (1):
- Miami Cancer Institute at Baptist Health, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Miami Cancer Institute website — http://baptisthealth.net/cancer-care/home

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Durvalumab Plus Radiation Therapy
Started | 9
Completed | 7
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Durvalumab Plus Radiation Therapy
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [66 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Time from initiation of durvalumab to progression per RECIST 1.1 or death, whichever comes first. Per RECIST 1.1, progressive disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions compared to baseline sum of target lesions, or any new lesions. Confirmation of PD for participants who are deemed clinically stable by the Investigator should be acquired preferably at the next regularly scheduled imaging visit and no earlier than 4 weeks after the prior assessment of PD.
Time Frame: 1 year
Population: Only 7 participants received study treatment. One participant voluntarily withdrew after signing consent, and one participant was a screen failure.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Durvalumab Plus Radiation Therapy
Number analyzed (Participants) | 7
days | 53 [51 to 53.5]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of the patients who have a complete response (CR) or partial response (PR) as defined by RECIST 1.1. The patient's best overall response rate defined as the best response recorded from the start of the treatment until disease progression. Per RECIST 1.1, CR is defined as the disappearance of all target lesions; PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. CR and PR requires a confirmatory scan preferably at the next regularly scheduled imaging visit and no earlier than 4 weeks after the prior assessment of CR, PR, or stable disease (SD).
Time Frame: 1 year
Population: Only 7 participants received study treatment. One participant voluntarily withdrew after signing consent, and one participant was a screen failure. An additional participant expired before their first follow-up imaging, so response could not be determined.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab Plus Radiation Therapy
Number analyzed (Participants) | 6
Participants | 0

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: The clinical benefit rate is the percentage of patients that have achieved a CR, PR, or stable disease (SD) as defined by RECIST 1.1. Per RECIST 1.1, CR is defined as the disappearance of all target lesions; PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters; PD is defined as at least a 20% increase in the sum of the diameters of target lesions compared to baseline sum of target lesions, or any new lesions; SD is defined as not meeting criteria for CR, PR, or SD. CR and PR requires a confirmatory scan preferably at the next regularly scheduled imaging visit and no earlier than 4 weeks after the prior assessment of CR, PR, or stable disease (SD). Confirmation of PD for participants who are deemed clinically stable by the Investigator should be acquired preferably at the next regularly scheduled imaging visit and no earlier than 4 weeks after the prior assessment of PD.
Time Frame: 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab Plus Radiation Therapy
Number analyzed (Participants) | 6
Participants | 1

4. Secondary Outcome: Time to In-field Progression
Description: In-field progression is defined as PD according to RECIST 1.1 criteria (at least a 20% increase in the sum of the diameters of target lesions compared to baseline sum of target lesions, or any new lesions) within the original field or area where the participant had been treated with radiation therapy. Confirmation of PD for participants who are deemed clinically stable by the Investigator should be acquired preferably at the next regularly scheduled imaging visit and no earlier than 4 weeks after the prior assessment of PD.
  The time to in-field progression is defined as the time from initiation of treatment to progression within the radiation.
Time Frame: 1 year
Population: Only 7 participants received study treatment; 3 participants demonstrated in-field progression.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Durvalumab Plus Radiation Therapy
Number analyzed (Participants) | 3
days | 53 [51 to 53.5]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first treatment until death. Patients who are alive will be censored at the last date of patient contact.
Time Frame: 1 year
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Durvalumab Plus Radiation Therapy
Number analyzed (Participants) | 7
days | 85 [75 to 175]

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Arm/Group | Durvalumab Plus Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 7/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab Plus Radiation Therapy (N=7)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Acute cystitis (Renal and urinary disorders) | 1 (1)
Rectal bleed (Gastrointestinal disorders) | 1 (1)
GI bleed (Gastrointestinal disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab Plus Radiation Therapy (N=7)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Increased alkaline phosphatase (Hepatobiliary disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Elevated troponin (Cardiac disorders) | 1 (1)
Generalized weakness (General disorders) | 1 (1)
Protein calorie malnutrition (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (3)
Low Albumin on Blood (Hepatobiliary disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Hyponatremia (Renal and urinary disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilateral pulmonary embolism (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early because of poor enrollment and participants being withdrawn soon after enrollment due to disease progression. Statistical analysis was not possible with the small number of evaluable participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03490760/Prot_SAP_000.pdf